CLINICAL TRIAL: NCT05093777
Title: Evaluation of a Norwegian Model of an Intensive Habilitation Program for Young Children With Early Brain Damage - a Multicentre Randomized Controlled Trial.
Brief Title: Program Intensive Habilitation (PIH) for Young Children With Early Brain Damage
Acronym: PIHMulti
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Jon Skranes, Professor dr med, Sorlandet Hospital HF
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KlinBeForskSkranes
Record Dates: First submitted 2021-09-28; First posted 2021-10-26 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Brain Injuries; Cerebral Palsy; Motor Skills Disorders; Empowerment; Parent-Child Relations; Parenting
Keywords: brain injury; cerebral palsy; motor disability; GMFCS level; Pedi-Cat; Family Empowerment scale; Parenting stress index
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy; Motor Skills Disorders; Empowerment | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT) with blinded evaluation by independent researchers at baseline, at 12 months and at 24 months. A stepped-wedge design will be applied so that all study participants eventually will be offered the intervention program. Those who are randomized to control group in the first year of study, will be offered intensive training during the second year, and vice versa.
Who Masked: Outcomes Assessor
Masking Description: Blinded evaluation by independent researchers at baseline, at 12 months and at 24 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Half of the study participants will be randomized to the intensive habilitation program the first year of program. The second year of program this group of participants will be offered habilitation "as usual".
  Interventions: Other: Program Intensified Habilitation; Other: Habilitation as usual
- Control group (Other): Half of the study participants will be randomized to "treatment as usual" the first year of program, then offered the intensive program during the second year ("stepped wedge design").
  Interventions: Other: Program Intensified Habilitation; Other: Habilitation as usual

INTERVENTIONS:
Other: Program Intensified Habilitation — The program is based on a holistic and family-centered concept, which acknowledges parents as experts on their child's abilities and needs. The program involves both parents and local professionals, and includes goal setting and goal-directed treatment targeted to the needs of the individual child. The program lasts for about one year and contains three in-patient group sessions over 2 weeks. In between the children are receiving individualized home training programs at home and in pre-school/kindergarten. The children train on a daily basis, both during the inpatient sessions and in the home setting.
  Other Names: PIH Multi
Other: Habilitation as usual — When the participants are not joining the study year containing the intervention program, they will be offered habilitation services "as usual" administered by the primary health care services in the local community.
  Other Names: Control

SUMMARY:
By longitudinal, prospective research in children with neurodisabilities including severe motor impairments and their parents to explore the beneficial effects of participating in an intensive habilitation program on the child's adaptive functioning and parental empowerment in order to treat and reduce the consequences of early brain damage.

DETAILED DESCRIPTION:
Evidence-based knowledge about the effects of intensive training programs for children with severe early brain damage is limited since research on this topic has methodological weaknesses and shows conflicting results. As intensive training programs require extensive efforts from the child, parents and professionals and represent major costs, the importance of scientifically proven effects is considerable. This research project aims to measure the effects of an intensive habilitation program for young children with severe early brain damage on the child's adaptive, motor, language and social functioning and on parental empowerment, family functioning and stress. In this randomized controlled trial (RCT) 90 children will be divided into an intervention group participating in a Norwegian developed program of intensified habilitation of 12 months duration and a control group, who will receive "services as usual" during the same time period. Between-group analyses will then be performed. Due to a stepped wedge design, the control participants will then be offered training in year two of participation. Within-group analysis of results before and after training will then be performed for all participants. Standardized measures with high responsiveness in documenting intervention effectiveness will be used as primary outcome measures. Intensive training groups will be offered in all Health Regions in Norway and if successful be implemented as standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* age 2 - 6 years at the start of the program
* a diagnosis of severe cerebral palsy or similar motor disability of non-progressive etiology (GMFCS level IV-V),
* being able to participate in group sessions
* having parents who want to take an active part in their child's training
* least one of the parents must speak fluent Norwegian or English.

Exclusion Criteria:

* children with progressive disorders
* co-morbidity like autism spectrum disorder, severe visual and hearing impairments or intractable epilepsy that worsen with physical activity.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Evaluation of Disability Inventory - Computer Adaptive Test (PEDI-CAT) | Change from baseline measure at 12 months and after 24 months
  Primary evaluation measure for the child
Change in Family Empowerment Scale (FES) | Change from baseline measure at12 months and after 24 months
  Primary evaluation measure for the parents

SECONDARY OUTCOMES:
Change in Gross motor function measure (GMFM-88) | Change from baseline measure at 12 months and after 24 months
  Secondary evaluation measure for the child
Change in Parenting Stress Index (PSI) | Change from baseline measure at 12 months and after 24 months
  Secondary evaluation measure for the parents

CONTACTS AND LOCATIONS:
Overall Officials: Jon Skranes, Principal Investigator — Sørlandet Hospital
Locations (1):
- Sørlandet Hospital, Kristiansand, Norway

IPD SHARING:
Plan to Share IPD: No